CLINICAL TRIAL: NCT06610955
Title: Effects of High Intensity Interval Training vs. Moderate Intensity Continuous Training on Fat Loss,Serum Adiponectin,Leptin,Omentin Level,Sleep and Quality of Life in Young Females With Obesity
Brief Title: Comparison of Two Different Intensity Exercises on Young Women With Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Collaborators: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Figen Tuncay, Professor, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AEU-FTR-EK-01
Record Dates: First submitted 2024-09-15; First posted 2024-09-24 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Exercise Training
Keywords: Obesity; Exercise Training; Adipokines
MeSH Terms: conditions — Obesity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Two groups without control group
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessments will be performed by a doctor who will be blinded to exercise group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity interval training exercise group (Active Comparator): After a 10 minutes warm up exercise, participants will exercise with a bicycle ergometry device at 80% of their maximum heart rate for 4 minutes, and the active recovery period will be 3 minutes (4x4 minutes). During the recovery period, the participant will exercise with the Ergoline bicycle ergometry system for 4 sets at 60% of their maximum heart rate for 3 minutes. A total of 45 minutes exercise session will be completed with a 10 minutes cool down exercise. Exercise will be done 5 days a week for a total of 8 weeks. In the first 4 weeks, exercise will be done at 80% intensity, and in the following weeks, the exercise intensity will be increased by 5% each week, respectively, to 85%, 90%, 95%, and 100% in the last week.
  Interventions: Other: High intensity interval training
- Moderate intensity continuous exercise group (Active Comparator): Following a 10 minutes warm up exercise, participants will exercise continuously for 30 minutes at 65% of their maximum heart rate with the Ergoline bicycle ergometry system. A 5 minutes cool down exercise will end the 45 minutes exercise session. The exercise duration is 5 days a week for a total of 8 weeks.
  Interventions: Other: Moderate intensity continuous training

INTERVENTIONS:
Other: High intensity interval training — After a 10 minutes warm up exercise, participants will exercise with a bicycle ergometry device at 80% of their maximum heart rate for 4 minutes, and the active recovery period will be 3 minutes (4x4 minutes). During the recovery period, the participant will exercise with the Ergoline bicycle ergometry system for 4 sets at 60% of their maximum heart rate for 3 minutes. A total of 45 minutes exercise session will be completed with a 10 minutes cool down exercise. Exercise will be done 5 days a week for a total of 8 weeks. In the first 4 weeks, exercise will be done at 80% intensity, and in the following weeks, the exercise intensity will be increased by 5% each week, respectively, to 85%, 90%, 95%, and 100% in the last week.
  Arms: High intensity interval training exercise group
Other: Moderate intensity continuous training — Following a 10 minutes warm up exercise, participants will exercise continuously for 30 minutes at 65% of their maximum heart rate with the Ergoline bicycle ergometry system. A 5 minutes cool down exercise will end the 45 minutes exercise session. The exercise duration is 5 days a week for a total of 8 weeks.
  Arms: Moderate intensity continuous exercise group

SUMMARY:
Obesity is one of the most common preventable public health problems. Diet regulation and exercise practices are the most commonly used methods in reducing fat tissue. There are various exercise methods applied in the weight loss process and the effects of different types of exercise modalities on body fat rate and metabolic status.The aim of our study is to determine the effects of high intensity interval exercise and moderate intensity continuous exercise on serum , omentin, leptin and adiponectin levels, anthropometric measurements used in obesity follow up, body fat percentage and their effects on the quality of sleep and life of women with obesity.

DETAILED DESCRIPTION:
Female participants aged 18-45 with a body mass index of 30-40 kg/m² who met the inclusion and exclusion criteria were randomized into two groups using a simple randomization method using a computer. One group will perform high intensity interval exercise with an Ergoline bicycle ergometry device for 45 minutes a day, 5 days a week for 8 weeks, while the other group will perform moderate intensity continuous exercise on the same device. Peripheral venous blood samples will be taken from all participants at the beginning and end of the study, anthropometric measurements used in obesity monitoring of all participants will be taken and noted, and participants will be asked to fill out questionnaires containing questions about their sleep and quality of life. The analysis of the blood samples taken will be carried out in the Biochemistry Laboratory of Kırşehir Ahi Evran University. The data of our study will be analyzed with the statistical package program SPSS version 23.0.

ELIGIBILITY:
Inclusion Criteria:

* Female between the age of 18-45
* BMI 30-40 kg/m²
* Primary obesity

Exclusion Criteria:

* Patients with cardiac, pulmonary, endocrinological, rheumatological diseases
* Pregnancy and breastfeeding
* Using antipsychotics, antidepressants (lithium, tricyclic antidepressants, mono amino oxidase inhibitors), anticonvulsants, antihistamines, glucocorticoids, antidiabetics (sulfonylureas, insulins, glitazones) sex hormones
* Using oral contraceptives
* History of bariatric surgery
* Patients using obesity medication in the last 6 months, complying with a regular diet and exercise program
* Presence of orthopedic or neurological problems that difficulty of participate aerobic exercise training

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Serum adipokine levels | 8 weeks
  This study aimed to investigate the effects of high intensity interval exercise and moderate intensity continuous exercise on serum adiponectin, leptin and omentin levels in young women with obesity.

SECONDARY OUTCOMES:
Anthropometric measurement | 8 weeks
  waist and hip circumference measurements
Percentage of body fat | 8 weeks
  skinfold thickness will measure with skinfold caliper
The impact of weight on quality of life | 8 weeks
  The impact of weight on quality of life will describe with The Impact of Weight on Quality of Life-Lite index
Quality of sleep | 8 weeks
  Sleep quality will describe Pittsburgh sleep quality index

CONTACTS AND LOCATIONS:
Overall Officials: Figen Tuncay, Professor, Principal Investigator — Ahi Evran Univeristy; Elif Kapaklı, RA, Study Chair — Kirsehir Ahi Evran Universitesi; Gamze Turna Saltoğlu, Ass. Prof., Study Chair — Kirsehir Ahi Evran Universitesi; Başak Çiğdem Karaçay, Assoc. Prof., Study Chair — Kirsehir Ahi Evran Universitesi; Nazife Kapan, Ass. Prof., Study Chair — Kirsehir Ahi Evran Universitesi; Başak Kavalcı Kol, Ass. Prof., Study Chair — Kirsehir Ahi Evran Universitesi; Merve Fırat, Ass. Prof., Study Chair — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran Üniversitesi, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Effect of High-Intensity Interval Training on Plasma Omentin-1 Concentration in Overweight/Obese and Normal-Weight Youth — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC5644954/